CLINICAL TRIAL: NCT05447416
Title: Intermittent Hypoxic Training (IHT) Versus Hyperbaric Oxygen Therapy (HBOT) for Aerobic Performance - Prospective Randomized Study
Brief Title: Intermittent Hypoxic Training (IHT) Versus Hyperbaric Oxygen Therapy (HBOT) for Aerobic Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Shay Efrati, MD, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 032-20-ASF
Record Dates: First submitted 2022-07-03; First posted 2022-07-07 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Healthy Active Athletes
Keywords: triathletes; cyclists; mitochondria; HBOT; HBO; IHT
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trail 2 groups treatment - HBOT and IHT
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperbaric Oxygen Therapy - HBOT (Active Comparator): The protocol comprises of 40 consecutive hyperbaric oxygen treatment (HBOT) sessions, 5 sessions per week within a two months' period. The HBOT group will train for 60 minutes after the HBOT sessions, 3 times per week, in a normobaric normoxic environment according to individualized training protocol
  Interventions: Device: Hyperbaric Oxygen Therapy - HBOT
- Intermittent Hypoxic Training - IHT (Active Comparator): The protocol comprises of 24 consecutive Intermittent Hypoxic Training (IHT) sessions, 3 sessions per week within a two months' period. Subjects will train according to individualized training protocol.
  Interventions: Device: Intermittent Hypoxic Training - IHT

INTERVENTIONS:
Device: Hyperbaric Oxygen Therapy - HBOT — Each session will include exposure of 90 minutes to 100% at 2 ATA, with 5 minutes air breaks every 20 minutes
  Arms: Hyperbaric Oxygen Therapy - HBOT
Device: Intermittent Hypoxic Training - IHT — Each session lasts 60 minutes of 15.2% oxygen at 1.0 ATA. Subjects will be training according to individualized training protocol.
  Arms: Intermittent Hypoxic Training - IHT

SUMMARY:
Comparing the effect of HBOT and IHT on aerobic performance of athletes.

DETAILED DESCRIPTION:
Enhanced physical performance is the goal of all professional and non-professional athletes. There are many intervention methods aim to enhance physical performance from 2 intervention related to change in the environment partial oxygen pressure have been demonstrated to have beneficial effect: IHT and HBOT.

This study offers one of the two interventions to athletes with a pre and post intervention objective evaluation of the physiological performance - Maximal exercise test for evaluating VO2MAX and ventilatory thresholds, time to exhaustion, 30 seconds Wingate test, agility test, muscle biopsy, blood tests, brain MRI, cognitive tests and exercise cognitive test.

After signing an informed consent form, eligible subjects will be randomized to one of the study groups at a ratio of 1:1. The IHT group will receive three hypoxic guided training sessions per week, according an individualized training protocol, 24 sessions in total.

The HBOT group will receive 40 daily hyperbaric sessions, five days per week. Each session will include 90 minutes exposure to 100% oxygen at 2ATA with a five-minute air break every 20 minutes. Three times per week, as the IHT group, the HBOT group will have a guided training session, according an individualized training protocol.

Both groups, IHT and HBOT, will have the same relative intensity guided training protocols for 8 weeks, to stimulate the same exercise load. The IHT group will train for 60 minutes, 3 times a week in a normobaric hypoxia environment, at O2 concentration of 15.2% that stimulates a 2500-2600m height. The HBOT group will train for 60 minutes after the HBOT sessions, 3 times per week, in a normobaric normoxic environment

Physical performance evaluations will be conducted on 3 different times post interventions - a day last intervention, 3 weeks after and 2 months after - in order to analyze the long term effect of each intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Vo2max above 3500 ml or Vo2max/kg above 50 ml/kg
2. Age 18-45
3. Subjects are active aerobic athletes, training regularly more than 4 exercise sessions per week.
4. Subject willing and able to read, understand and sign an informed consent

Exclusion Criteria:

1. Inability to attend scheduled clinic visits and/or comply with the study protocol
2. Active malignancy
3. Active smokers
4. Previous treatment of HBOT for any reason prior to study enrollment.
5. Chest pathology incompatible with pressure changes
6. Major orthopedic injury at the past 3 months
7. Inner ear disease
8. Lung pathology
9. The inability to perform an awake brain MRI
10. Claustrophobia
11. Previous neurologic conditions (e.g., Epilepsy, Brain tumors or s/p neurosurgery etc.)
12. Comorbidities and medications that rule out the subject

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male biologically
Enrollment: 66 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary exercise test (CPET) | Baseline, 11 weeks
  CPET determines the gas exchange dynamics that is expected to change through the intervention

SECONDARY OUTCOMES:
Cardiopulmonary exercise test (CPET) | 8 weeks, 16 weeks
  CPET determines the gas exchange dynamics that is expected to change through the intervention
Time To Exhaustion | Baseline, 11 weeks, 16 weeks
  The test will be conducted on the SRM high performance ergometer on 105% of the maximal aerobic power
Wingate 30 seconds anaerobic test | Baseline, 11 weeks, 16 weeks
  The Wingate Anaerobic Test (WAnT) is conducted on the SRM high performance ergometer.
Muscle biopsy for mitochondrial function | Baseline, 11 weeks
  Participants will undergo a muscle biopsy, muscle sample will be analyzed using the Oxygraph (Oroboros Inc, Austria) for oxygen respiratory function, as well as staining for mitochondrial proteins
Blood test for evaluation of CBC | Baseline, 11 weeks, 16 weeks
  complete blood count
Blood test for evaluation of HIF-1α | Baseline, 7 weeks, 8 weeks, 11 weeks, 16 weeks
  Hypoxic inducible factor 1α levels
Blood test for evaluation of Telomeres length | Baseline,11 weeks, 16 weeks
  Using staining and FACS technology telomere length will be analyzed
Blood test for evaluation of mitochondrial function | Baseline,11 weeks
  Mitochondrial function of Peripheral Blood Mononuclear Cells (PBMC) and Platelets (PLT)

OTHER OUTCOMES:
Cognitive Function | Baseline, 11 weeks
  Cognitive function will be evaluated using the Neurotrax computerized cognitive assessment and the Cambridge Neuropsychological Test Automated Battery (CANTAB).
Cognitive Function under exercise | Baseline, 11 weeks
  Participants will be asked to pedal on a bike on workload correlated to 85% of the second ventilatory threshold obtained during the CPET and will simultaneously perform a Stroop test using the EncephalApp Stroop Test application on a tablet.
Whole-brain quantitative perfusion imaging | Baseline, 11 weeks
  Whole-brain quantitative perfusion imaging will be performed using Dynamic susceptibility contrast (DSC)-MRI technique
Brain microstructure MRI evaluation | Baseline, 11 weeks
  Fractional anisotropy (FA) and Mean diffusivity (MD) will be evaluated using diffusion tensor imaging (DTI) MRI protocol
Brain functional connectivity imaging | Baseline, 11 weeks
  Resting state functional MRI
Pulse Rate variability and activity | baseline to 16 weeks
  Participants will be asked to wear a smartwatch (Garmin, USA) in the entire time frame of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Shai a Efrati, MD, Principal Investigator — Asaf-Harofhe MC
Locations (1):
- The Sagol Center for Hyperbaric Medicine and Research Shamir Medical Center (Assaf Harofeh), Zrifin, Israel

IPD SHARING:
Plan to Share IPD: No